CLINICAL TRIAL: NCT05730413
Title: Once Versus Twice Bisoprolol Dosage Regimen in Prevention of Atrial Fibrillation Post Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Ihab Farouq, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CL(2776)
Record Dates: First submitted 2023-01-27; First posted 2023-02-15 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Bypass Grafting; Postoperative Atrial Fibrillation; Coronary Artery Disease
Keywords: Bisoprolol; Dosage regimens; heart rate; blood pressure
MeSH Terms: conditions — Coronary Artery Disease | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Once Daily Regimen (Active Comparator): Patients who take bisoprolol 5 mg per day.
  Interventions: Drug: Bisoprolol
- Twice Daily Regimen (Experimental): Patients who take bisoprolol 2.5 mg twice per day.
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol dose was divided to be taken as 2.5 mg twice per day from hospital admission to discharge.
  Arms: Twice Daily Regimen
Drug: Bisoprolol — Bisoprolol was taken as 5 mg per day from hospital admission till discharge.
  Arms: Once Daily Regimen

SUMMARY:
The goal of this interventional clinical trial is compare between two different dose regimens of bisoprolol (beta-blocker) in CABG patients in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients: 18 to 65 years old
* Diagnosed with coronary heart disease or myocardial infarction and scheduled for coronary artery bypass surgery

Exclusion Criteria:

* History of Ventricular arrhythmia, atrial fibrillation, atrial flutter, left bundle block, AV block grade II/III
* History of Sick sinus syndrome, sinoatrial heart block
* History of valve replacement
* Permanent Pacemaker
* LVEF less than 30%
* Unstable Heart failure
* Cardiogenic shock
* Sustained systolic blood pressure less than 100 mmHg or HR less than 50 bpm at recruitment
* Severe chronic obstructive airway disease
* Severe asthma unless was on previously tolerated bisoprolol dose
* Uncontrolled diabetes mellitus unless was on previously tolerated bisoprolol dose
* Pregnant/Lactation
* Previous recent stroke
* Creatinine clearance less than 30 ml/min
* End stage liver disease (liver cirrhosis)
* Drug dependance history
* Untreated phaeochromocytoma
* Vasospastic angina
* Thyrotoxicosis
* History of advanced staged of peripheral vascular disease
* Hypersensitivity
* Patients on any other beta-blocker other than bisoprolol
* Patients on bisoprolol higher than 5 mg/day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Prevention of postoperative Atrial fibrillation without normal blood pressure and/or heart rate | 5 days
  Incidence of Atrial Fibrillation

SECONDARY OUTCOMES:
Onset time of Atrial Fibrillation | 5 days
  Time at which event happened.
Recurrence of Atrial Fibrillation | 5 days
  Time at which event recurred.
Mean reduction in heart rate | Hospital stay ( up to 10 days)
  Mean of reduction between two arms.
Mean resting heart rate | Hospital stay ( up to 10 days)
  mean resting heart rate between two arms.
Mean systolic and diastolic blood pressure | Hospital stay (up to 10 days)
  Mean systolic and diastolic blood pressure between two arms.
Length of ICU stay | ICU stay (up to 5 days)
  time spent in the from ICU admission to ICU discharge
Length of Hospital stay | Hospital stay (up to 10 days)
  time spent in the hospital till discharge
Medication safety | Hospital stay (up to 10 days)
  Any symptom which requires dose lowering or discontinuation of bisoprolol e.g hypotension episodes
Bisoprolol concentration | time before next dose post average 24 hours
  Bisoprolol concentration between two arms
Use of inotropes/vasopressors | ICU stay (up to 5 days)
  compare use of inotropes/vasopressors between the two arms.
ICU mortality | ICU stay (up to 5 days)
  Number of death during ICU stay
Hospital Mortality | Hospital Stay (up to 10 days)
  Number of death during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Reem Ihab, Bsc, Principal Investigator — Cairo University
Locations (1):
- El-Demerdash Cardiac Academy Hospital, Cairo, Egypt